CLINICAL TRIAL: NCT03376152
Title: Rural China Electric Kettle Promotion Program: a Cluster-Randomized Controlled Trial of Pilot Program Impact on Electric Kettle Adoption, Drinking Water Quality, Indoor Air Pollution, and Reported Health Outcomes in Poverty Households in the People's Republic of China
Brief Title: Rural China Electric Kettle Promotion Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Center for Rural Water Supply Technical Guidance (NCRWSTG), China (Unknown); Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Alasdair Cohen, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016119356
Record Dates: First submitted 2017-11-28; First posted 2017-12-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Compliant Behavior; Diarrheal Disease; Pollution; Exposure
MeSH Terms: conditions — Cooperative Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Active Comparator): "Poverty households" invited to attend cluster-level electric kettle promotion events and offered free kettles, information, and promotional materials 450 households in 15 clusters (30 households per cluster)
  Interventions: Behavioral: Electric Kettle Promotion
- Control Arm (No Intervention): 450 households in 15 clusters (30 households per cluster)

INTERVENTIONS:
Behavioral: Electric Kettle Promotion — Provision of free electric kettles and promotional materials/information
  Arms: Treatment Arm

SUMMARY:
This study will evaluate the impact of a pilot Rural Electric Kettle Promotion Program offered to low-income households in rural Anhui Province, China. The primary objective of this study is to determine whether this promotion program causes poverty households currently boiling their drinking water with solid-fuels (or drinking untreated water or bottled water) to switch to boiling their drinking water with electric kettles, and if so, how such a switch might improve safe drinking water access and/or reduce household air pollution.

DETAILED DESCRIPTION:
Previous research suggests that increasing the use of electric kettles for boiling (i.e., treating) drinking water in low-income areas of rural China could help expand access to safer drinking water, reduce household air pollution, and improve environmental and health outcomes in rural Chinese households currently boiling drinking water with solid-fuels (or not treating their water, or drinking contaminated bottled water).

The study will use a parallel arm cohort cluster-randomized controlled trial design with a 1:1 ratio. The study will randomize 30 clusters (i.e., villages) to treatment or control using stratified randomization by geography (two levels: mountains and plains) and by cluster proportions of reported electric kettle use at baseline. Randomization sequence generation will be conducted by A. Cohen using a random number generator (with a reproducible seed) in Stata v.13.1 (StataCorp, College Station, Texas, USA).

The study will collect data from 30 randomly selected households in 15 villages, for a total of 900 households. This sample size was powered to measure a 15% (or larger) change in electric kettle adoption, because the Chinese Center for Disease Control and Prevention (China CDC) will be unlikely to rollout a national program if adoption rates are less than 15%.

After baseline data collection and randomized allocation, in the intervention group village-level promotion events will take place in November-December of 2017, and will be organized by the provincial and county China CDC, in collaboration with the National Center for Rural Water Supply Technical Guidance (NCRWSTG). At these promotion events, households in the intervention group will be provided free, food-grade quality, electric kettles, as well as promotional materials (a calendar and poster) and information about the benefits of electric kettle use and improved hygiene and sanitation practices.

Because of known issues with decreasing adoption of drinking water treatment after behavior change promotion interventions such as this, and considering expected seasonal variation in boiling practices and frequencies, study data was initially planned to be collected over a period of 12 months (with additional qualitative follow-up via focus groups: 2019-03, 2019-08).

We were able to extend the follow-up data collection period from 12-months to 24-months, so we did not collect data from focus groups in 2019-03 or 2019-08 as originally planned. Follow-up data collection was completed in November 2019.

Due to the COVID-19 pandemic, we again postponed plans to collect data from focus groups (data cleaning efforts were delayed until 2021, and completed at the end of 2022). Logistics allowing, we hope to collect data from focus groups in 2023.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 18 or older will be eligible to provide consent for their households.
* Government classified "poverty households" (poverty classification based on 2016 data/records).

Exclusion Criteria:

* Persons aged 17 or younger will not be eligible to provide consent for their households.
* We will not have any exclusion criterion based on gender, race, ethnicity, language, or literacy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2017-11-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of households using electric kettles for boiling drinking water | 24 months.
  Primary measurement via electricity use meters (Tepsung model 10/16A) affixed to electric kettle power cables for all household who report using electric kettles at each of five visits (based on total KWh consumed per data collection intervals and estimated mean liters boiled per person, per day, per household, by electric kettle type/size). Additional measurement via self-report of electric kettle use (household surveys) and via enumerator direct observations (during visits to households).

SECONDARY OUTCOMES:
Thermotolerant coliforms in household point-of-consumption drinking water | 6 months.
  Point-of-consumption drinking water sample collection from subsample of households (150 in each arm, 300 total) and laboratory analysis via multiple tube fermentation (using China CDC national standards and protocol) for Thermotolerant coliforms, an indicator of fecal contamination.
Diarrhea prevalence | 24 months.
  Self-report (current, 7-day recall, 14-day recall)
Particulate matter 2.5 mg/m3 (PM2.5) concentrations | 1 month.
  Custom-built air pollution sensors (PM2.5 and other - developed by Prof. Tao Shu et al. at Peking University, Beijing, CHINA) installed to collect indoor air pollution data for 3-4 weeks in a subsample of households (40-50 in each arm, 80-100 total), with 3-5 external air pollution sensors installed in each cluster to control for ambient air pollution.
Prevalence of hand washing with soap | 24 months.
  Self-report during household surveys combined with enumerator direct observations

OTHER OUTCOMES:
Cough prevalence | 24 months.
  Self-report (current, 7-day recall)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Tao, Director, Principal Investigator — National Center for Rural Water Supply Technical Guidance
Locations (1):
- National Center for Rural Water Supply Technical Guidance，Chinese Center for Disease Control and Prevention, Beijing, China

IPD SHARING:
Plan to Share IPD: No